CLINICAL TRIAL: NCT03236805
Title: Intravenous Subdissociative-dose Ketamine Versus Morphine for Prehospital Analgesia a Randomized Controlled Trial
Brief Title: Intravenous Subdissociative-dose Ketamine Versus Morphine for Prehospital Analgesia
Acronym: KETAMORPH
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: 285 patients have recruited instead on 496 but we don't want to continue to prolonge the study. Analysis will be performed on the data we have.
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC17_0082
Record Dates: First submitted 2017-07-17; First posted 2017-08-02 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Pain Management
Keywords: Morphine; Ketamine; Acute pain; prehospital
MeSH Terms: conditions — Agnosia; Acute Pain | interventions — Ketamine; Morphine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamine IV (Experimental)
  Interventions: Drug: Ketamine
- Morphine IV (Active Comparator)
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Ketamine — Initial bolus of 20 mg (around 0.3 mg per kg) followed by bolus of 10 mg every 5 minutes as reported by the recommandations of experts of the french society of urgency care
  Arms: Ketamine IV
Drug: Morphine — Bolus of 2 mg (patient with weight under 60 kgs) or bolus of 3 mg (patient with weight above 60 kgs) every 5 minutes as reported by the recommandations of experts of the french society of urgency care
  Arms: Morphine IV

SUMMARY:
This is a prospective, randomized, single-blind trial evaluating prehospital patients experiencing moderate to severe acute pain, defined as a numeric rating scale score greater than or equal to 5. Patients will be randomized to receive ketamine at or morphine by intravenous push.

DETAILED DESCRIPTION:
This study is designed to evaluate if ketamine alone is non inferior to morphine alone for prehospital analgesia. Numeric rating scale pain scores will be compared between recipients of ketamine and recipients of morphine at 15, 30, 45 and 60 min post first injection and at hospital admission.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years old
* prehospital moderate to severe acute pain, defined as a numeric rating scale score greater than or equal to 5

Exclusion Criteria:

* unstable vital signs (systolic blood pressure <90 or >200 mm Hg, pulse rate <50 or >150 beats/min, and respiration rate <10 or >30 breaths/min)
* pregnancy
* breast-feeding
* altered mental status
* unable to give numeric rating scale scores
* allergy to morphine or ketamine
* acute pulmonary edema
* acute coronary syndrome
* renal or hepatic insufficiency
* patient who received morphine for the same acute pain
* acute psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2017-11-23 (Actual); Primary Completion 2022-11-26 (Actual); Study Completion 2022-11-26 (Actual)

PRIMARY OUTCOMES:
Comparison of numeric rating scale pain scores between recipients of ketamine and morphine at 30 minutes post first injection. | 30 minutes

SECONDARY OUTCOMES:
Comparison of numeric rating scale pain scores between recipients of ketamine and morphine at 15 minutes post first injection. | 15 minutes
Comparison of numeric rating scale pain scores between recipients of ketamine and morphine at 45 minutes post first injection. | 45 minutes
Comparison of numeric rating scale pain scores between recipients of ketamine and morphine at 60 minutes post first injection. | 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Joel JENVRIN, Doctor, Principal Investigator — Nantes University Hospital
Locations (12):
- France (12):
  - Angers University Hospital, Angers
  - University Hospital of Bordeaux, Bordeaux
  - Hospital of Chateaubriant, Châteaubriant
  - CH de Gonesse, Gonesse
  - Grenoble University Hospital, Grenoble
  - La Roche sur Yon Hospital, La Roche-sur-Yon
  - Le Mans University Hospital, Le Mans
  - Nantes University Hospital, Nantes
  - Quimper Hospital, Quimper
  - Rennes University Hospital, Rennes
  - Hospital of Saint Nazaire, Saint-Nazaire
  - Tours University Hospital, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Le Cornec C, Le Pottier M, Broch H, Marguinaud Tixier A, Rousseau E, Laribi S, Janiere C, Brenckmann V, Guillerm A, Deciron F, Kabbaj A, Jenvrin J, Pere M, Montassier E. Ketamine Compared With Morphine for Out-of-Hospital Analgesia for Patients With Traumatic Pain: A Randomized Clinical Trial. JAMA Netw Open. 2024 Jan 2;7(1):e2352844. doi: 10.1001/jamanetworkopen.2023.52844. PMID 38285446
- [Derived] Le Cornec C, Lariby S, Brenckmann V, Hardouin JB, Ecoffey C, Le Pottier M, Fradin P, Broch H, Kabbaj A, Auffret Y, Deciron F, Longo C, Javaudin F, Le Bastard Q, Jenvrin J, Montassier E. Is intravenously administered, subdissociative-dose KETAmine non-inferior to MORPHine for prehospital analgesia (the KETAMORPH study): study protocol for a randomized controlled trial. Trials. 2018 May 2;19(1):260. doi: 10.1186/s13063-018-2634-3. PMID 29716637